CLINICAL TRIAL: NCT02260661
Title: A Phase I, Open-Label, Multicentre, Dose-Escalation Study to Investigate the Safety and Pharmacokinetics of AZD8835 in Patients With Advanced Solid Tumours
Brief Title: Phase I, Dose Study to Look at the Safety and Pharmacokinetics of AZD8835 in Patients With Advanced Solid Tumours
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D6140C00001
Record Dates: First submitted 2014-10-06; First posted 2014-10-09 (Estimated); Last update posted 2016-10-10 (Estimated); Status verified 2016-10

CONDITIONS: Advanced Solid Malignancies; Breast Cancer - ER+, HER2 -; Breast Cancer - ER+, HER2-, PIK3CA Gene Mutation
Keywords: AZD8835; Fulvestrant; Breast Cancer; PIK3CA Gene Mutation
MeSH Terms: conditions — Breast Neoplasms | interventions — AZD8835; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Part A (Experimental): AZD8835 single agent dose escalation
  Interventions: Drug: AZD8835
- Part B (Experimental): Following the single agent dose escalation (Part A), additional patients with mutations in the PIK3CA gene will be enrolled to a single agent dose expansion phase at the MTD or recommended phase II dose (RP2D) at the selected dose schedule (as appropriate) to explore further the safety, tolerability, pharmacokinetics and biological activity at the selected dose (Part B). Part B will include patients with ER+/HER2 negative breast cancer whose tumours have a mutation of the PIK3CA gene and patients with any solid tumours which have a mutation of the PIK3CA gene.
  Interventions: Drug: AZD8835
- Part C (Experimental): AZD8835 in combination with fulvestrant dose escalation
  Interventions: Drug: AZD8835 in combination with fulvestrant
- Part D (Experimental): Following the combination dose escalation segment of the study (Part C), additional postmenopausal patients with ER+/HER negative breast cancer and mutations of the PIK3CA gene will be enrolled to a AZD8835 and fulvestrant combination dose expansion phase at the maximum tolerated dose (MTD) or recommended phase II dose (RP2D) (as appropriate) to explore further the safety, tolerability, pharmacokinetics and biological activity at the selected dose (Part D).
  Interventions: Drug: AZD8835 in combination with fulvestrant

INTERVENTIONS:
Drug: AZD8835 — AZD8835 is a small molecule that inhibits cancer progression by blocking PI3 kinase pathway components
  Arms: Part A
Drug: AZD8835 — AZD 8835 is a small molecule that inhibits cancer progression by blocking PI3 kinase pathway components
  Arms: Part B
Drug: AZD8835 in combination with fulvestrant — AZD8835 is a small molecule that inhibits cancer progression by blocking PI3 kinase pathway components. Fulvestrant is approved for the treatment of postmenopausal women with ER+ locally advanced or metastatic breast cancer following progression of disease while receiving anti-estrogen therapy.
  Other Names: Faslodex
  Arms: Part C
Drug: AZD8835 in combination with fulvestrant — AZD8835 is a small molecule that inhibits cancer progression by blocking PI3 kinase pathway components. Fulvestrant is approved for the treatment of postmenopausal women with ER+ locally advanced or metastatic breast cancer following progression of disease while receiving anti-estrogen therapy
  Other Names: Faslodex
  Arms: Part D

SUMMARY:
First time in patients study of AZD8835. The study has four parts. Part A AZD8835 is administered as a single agent in a multiple ascending dose escalation phase to investigate dose level for monotherapy. Part B follows the multiple ascending dose phase, additional patients with tumors with documented PIK3CA gene mutation will be enrolled to a single dose expansion phase. Part C is a second dose escalation phase in which post-menopausal patients with estrogen receptor positive (ER+), HER2 negative breast cancer will receive AZD8835 in combination with fulvestrant. Part D follows the combination dose escalation phase of the study, additional postmenopausal patients with ER+/HER2 negative breast cancer with documented PIK3CA gene mutation will be enrolled to a AZD8835 and fulvestrant combination dose-expansion phase at maximum tolerated dose or recommended phase II dose.

DETAILED DESCRIPTION:
AZD8835 is a novel small molecule that inhibits cancer progression by blocking PI3 kinase pathway components p110α and p110δ.

In this first-time-in-patient study, AZD8835 will initially be administered as a single agent to patients with advanced solid malignancies. Patients will be treated at a starting dose of 20 mg twice daily (BID), administered weekly on Days 1 and 4 and will be escalated to reach a maximum-tolerated dose (MTD) in patients as defined by dose-limiting toxicities (DLTs). A BID intermittent dosing schedule administered weekly on Days 1 and 4 of an oral formulation of AZD8835 will be used, as deemed optimal and effective in non-clinical studies, primarily to determine the safety and tolerability of AZD8835. The pharmacokinetics (PK) of AZD8835 and potential biological activity will also be investigated. In Part A of this study, AZD8835 will be administered as a single agent in a multiple ascending dose escalation phase to investigate the appropriate monotherapy dose level for clinical use. Additional dosing schedules may be studies, including dosing on Days 1 and 2 of each week, rather than Days 1 and 4.

Backfilled pharmacodynamic (PDc) cohorts in selected patients with tumours that have documented mutations in the phosphatidylinositol-4,5- bisphosphate 3-kinase, catalytic subunit alpha (PIK3CA) gene will allow further preliminary assessment of the biological effect of AZD8835 in these patients.

Following the single-agent dose-escalation phase of the study, additional patients with tumours that have documented mutations in the PIK3CA gene will be enrolled to a single-agent dose-expansion phase at the MTD or recommended Phase II dose (RP2D) at the selected dose schedule (as appropriate) to explore further the safety, tolerability, PK, and biological activity at the selected dose (Part B).

In addition, a further dose-escalation phase will be initiated following the observation of specific pre-determined criteria in the single-agent dose escalation, in which postmenopausal patients with oestrogen receptor positive (ER+), HER2 negative breast cancer will receive AZD8835 in combination with fulvestrant (Part C). The combination dose-escalation phase will investigate the appropriate combination dose level for clinical use.

Following the combination dose-escalation phase of the study, additional postmenopausal patients with ER+ breast cancer and tumours with documented mutations of the PIK3CA gene will be enrolled to a AZD8835 and fulvestrant combination dose-expansion phase at the MTD or RP2D (as appropriate) to explore further the safety, tolerability, PK, and biological activity at the selected dose (Part D).

ELIGIBILITY:
Inclusion Criteria:

1. Part A: Histological or cytological confirmation of a solid tumor and disease progression. Part B: Histological or cytological confirmation of ER positive, HER2 negative breast cancer and disease progression or any other solid tumor with a PIK3CA gene mutation. Part C: Histological or cytological confirmation of ER positive, HER2 negative postmenopausal breast cancer with locally advanced or metastatic disease that is eligible for fulvestrant treatment. Part D: Histological or cytological confirmation of ER positive, HER2 negative postmenopausal breast cancer with locally advanced or metastatic disease that is eligible for fulvestrant treatment. Patients must also present with a tumor related mutation of the PIK3CA gene.
2. Availability of archival tumour tissue sample. If archival sample is not available, a fresh tumour biopsy must be provided.
3. At least one measurable lesion per RECIST v1.1. However, breast cancer patients with only bone disease are also eligible.
4. ECOG Performance Status 0-1.
5. Adequate organ function at baseline:

   1. Serum total bilirubin ≤ 1.5 x ULN and AST/SGOT and ALT/SGPT ≤ 2.5 x ULN or ≤ 5 x ULN if liver metastases are present.
   2. Creatinine ≤ 1.5 x ULN, or calculated or measured creatinine clearance ≥ 50 mL/min, or 24-hour measured urine creatinine clearance ≥ 50 mL/min.
   3. Platelets ≥ 100 x 10^9, Hb ≥ 90 g/L, ANC ≥ 1.5 x 10^9/L.
   4. aPTT ≤ 1.5 x ULN
   5. Fasting glucose < 140 mg/dL (7.8 mmol/L).
   6. Glycated haemoglobin (HbA1c) < 8%
6. Female patients and male patients with female partners of child bearing potential must be using adequate contraception.

Exclusion Criteria:

1. Recent chemotherapy, radiotherapy, hormonal therapy, immunotherapy or investigational drugs within 21 days or 5 half-days from enrolment.
2. Received palliative/focal radiotherapy within 2 weeks of first dose of study treatment.
3. Major surgery ≤ 21 days from beginning of study drug
4. Any of the following cardiac criteria: CHF > Class II, cardiac ventricular arrhythmia requiring therapy, unstable angina or new-onset angina, QTcF interval >470ms, abnormal ECHO or MUGA at baseline (LVEF <50%).
5. Leptomeningeal disease
6. Part A: Intolerable AEs due to other PI3K inhibitors, dual PI3K and mTOR inhibitors or AKT inhibitors. Parts B, C, and D: Prior exposure to any of the following: pharmacological inhibitors of AKT, PI3K, or dual PI3K and mTOR kinase activity
7. Strong inhibitors and potent inducers of CYP3A4
8. Peripheral neuropathy CTCAE v4.03 Grade ≥ 3
9. Diarrhoea CTCAE v4.03 Grade ≥ 2
10. Acute or chronic pancreatitis
11. Clinically manifest diabetes mellitus, history of gestational diabetes mellitus and/or known glucose intolerance.
12. Patients currently receiving any medication that has the potential to prolong the QT interval or induce Torsades de Pointes
13. Spinal cord compression or brain metastases unless asymptomatic and not requiring steroids for at least 4 weeks
14. Patients in the combination arms - known hypersensitivity to fulvestrant
15. Therapeutic treatment with Coumadin or any other coumarin-derivative anticoagulant
16. Impaired GI function or GI disease that may interfere with absorption of AZD8835 or patients unable to take oral medication
17. As judged by the investigator any evidence of severe or uncontrolled systemic disease
18. Patients treated with hematopoietic colony-stimulating growth factors e.g., G-CSF, GM-CSF, M-CSF) ≤ 2 weeks prior to start. Erythropoietin or darbepoetin is allowed if it was initiated at least 2 weeks prior to entry

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-11; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Determine the maximum tolerated dose (MTD) or recommended Phase II dose of oral AZD8835 as a single agent and in combination with fulvestrant | At the end of one cycle of treatment
  MTD - A dose will be considered non-tolerated and dose escalation will stop if 2 or more of up to 6 evaluable patients experience a dose limiting toxicity at a dose level. Once the non-tolerated dose is defined, the MTD will be confirmed at the previous dose level below the non-tolerated dose or a dose between the non-tolerated dose and the last tolerated dose my be investigated. A minimum of 6 evaluable patients are required to determine the MTD. Recommended Phase II dose - A minimum of 6 evaluable patients is necessary to determine the recommended dose. A dose will be considered non-tolerated and dose escalation will stop if 2 or more patients experience a dose dose limiting toxicity at a dose level.
Establish the preliminary safety and tolerability profile of oral AZD8835 as a single agent and in combination with fulvestrant | Up to a projected 36 months
  Assessed in terms of adverse events and laboratory data that is collected on all patients

SECONDARY OUTCOMES:
To establish the pharmacokinetic profile of oral AZD8835 as a single agent and in combination with fulvestrant | Venous blood samples will be collected pre-dose and at 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, and 96 hours post dose - exact schedule varies according to Part A, B, C, or D
  Venous blood samples (2 mL) for determination of concentrations of AZD8835 and the investigation of AZ8835 metabolites in plasma will be taken during Parts A, B, C, D
To evaluate the preliminary efficacy and anti-tumor activity of oral AZD8835 as a single agent or in combination with fulvestrant | Tumour response will be assessed at the completion of Cycle 2 (Week 8) and patients will be restaged after every 8 weeks for up to 1 year and every 12 weeks thereafter; assessments should be performed until disease progression.
  Categorization of objective tumor response will be based on RECIST v1.1 guidelines for complete response, partial response, stable disease, or progression of disease
To evaluate the pharmacodynamic (PDc) effect of oral AZD8835 as a single agent and in combination with fulvestrant | Tumour biopsies will be collected: (1) at pretreatment, (2) at one on-treatment time point (preferably Cycle 2 Day 1), and (3) at end of study treatment (preferably at disease progression)
  Tumor samples will be analyzed to assess PRAS40 phosphorylation, AKT phosphorylation, S6 phosphorylation, FOXO3a localisation

CONTACTS AND LOCATIONS:
Overall Officials: Hendrik-Tobias Arkenau, FRCP, PhD, Principal Investigator — Sarah Cannon Research Institute, United Kingdom
Locations (9):
- United States (5):
  - Research Site, Denver, Colorado
  - Research Site, Greenville, South Carolina
  - Research Site, Nashville, Tennessee
  - Research Site, Houston, Texas
  - Research Site, Milwaukee, Wisconsin
- United Kingdom (4):
  - Research Site, Cambridge
  - Sarah Cannon Research Institute, United Kingdom, London
  - Research Site, London
  - Research Site, Manchester